CLINICAL TRIAL: NCT00049582
Title: Phase I Study of 5-Aza-2'-Deoxycytidine (Decitabine) as a Biologic Modifier of Retinoid Responsive Genes in Patients With High-Risk Myelodysplastic Syndromes and Acute Myelogenous Leukemia (De-novo, Relapsed or Secondary)
Brief Title: Decitabine in Treating Patients With Myelodysplastic Syndromes or Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02502; NCI-2012-02502 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000258121; NCI-5591; PHL-004; PHL-004 (Other: Princess Margaret Hospital Phase 2 Consortium); 5591 (Other: CTEP); N01CM62203 (NIH)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; de Novo Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Leukemia, Myeloid, Acute | interventions — Decitabine

ARMS (1):
- Treatment (decitabine) (Experimental): Patients receive decitabine IV over 3 hours twice daily OR IV over 1 hour once daily on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of decitabine until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.
  Interventions: Drug: decitabine; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: decitabine — Given IV
  Other Names: 5-aza-dCyd; 5AZA; DAC
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of decitabine in treating patients with myelodysplastic syndromes or acute myeloid leukemia. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of decitabine in patients with high-risk myelodysplastic syndromes or acute myeloid leukemia.

II. Determine the minimum effective dose of this drug that produces demethylation of DNA with tolerable toxicity in these patients.

III. Determine the minimum effective dose of this drug that augments in vitro responses to retinoids.

IV. Determine the pharmacokinetics of this drug in these patients. V. Determine the clinical response rate of patients treated with this drug.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive decitabine IV over 3 hours twice daily OR IV over 1 hour once daily on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of decitabine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A maximum of 36 patients will be accrued for this study within 18 months.

ELIGIBILITY:
Inclusion Criteria:

* One of the following diagnoses:

  * High-risk myelodysplastic syndromes (MDS)
  * Acute myeloid leukemia (AML)

    * De novo, secondary, or relapsed disease
    * Any number of prior regimens for primary or relapsed disease
* Ineligible for or refuses aggressive management
* Measurable disease, defined as:

  * More than 5% blasts in bone marrow of patients with MDS
  * More than 30% blasts in bone marrow of patients with AML
* Involvement of cerebrospinal fluid allowed
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* See Disease Characteristics
* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* AST and/or ALT no greater than 1.25 times ULN
* Creatinine less than 1.7 mg/dL
* Creatinine clearance at least 60 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No ongoing or active infection
* No other uncontrolled illness that would preclude study participation
* No psychiatric illness or social situation that would preclude study compliance
* No prior allergic reactions to compounds of similar chemical or biological composition to decitabine
* No other active malignancy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* At least 4 weeks since prior biologic therapy (e.g., interferon, filgrastim [G-CSF], sargramostim [GM-CSF], thrombopoietin, or epoetin alfa)
* No concurrent hematopoietic growth factors (GM-CSF, thrombopoietin, or epoetin alfa)
* No concurrent prophylactic G-CSF
* Prior intrathecal cytarabine allowed for patients with cerebrospinal fluid involvement
* At least 4 weeks since prior chemotherapy (except low-dose chemotherapy administered to maintain WBC counts) (6 weeks for nitrosoureas or mitomycin) and recovered
* At least 24 hours since prior hydroxyurea
* Concurrent intrathecal cytarabine allowed for patients with cerebrospinal fluid involvement
* No prior radiotherapy greater than 3,000 cGy to marrow-producing areas
* At least 4 weeks since prior radiotherapy and recovered
* Prior investigational therapy allowed
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-09; Primary Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of decitabine, graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v2.0 | Up to day 28

SECONDARY OUTCOMES:
Minimal effective dose of decitabine that will lead to demethylation of deoxyribonucleic acid (DNA) with tolerable toxicity as assessed by RXR gene | Up to day 28
Proportion of patients with in-vitro retinoid response | Up to 8 years
Duration of clinical response | Up to 8 years
Changes in gene expression, gene methylation and bone marrow aspirate sample measurements | Up to day 5
  The effect on gene expression due to pharmacological exposures (ie retinoic acid receptor [RAR] or retinoid X receptor [RXR]) will be assessed using chi-square tests.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Minden, Principal Investigator — Princess Margaret Hospital Phase 2 Consortium
Locations (1):
- Princess Margaret Hospital Phase 2 Consortium, Toronto, Ontario, Canada